CLINICAL TRIAL: NCT04037852
Title: Robotic Versus Conventional or Endoscopic Nipple Sparing Mastectomy in the Management of Breast Cancer- A Prospective Registry Case Control Study
Brief Title: Robotic Versus Conventional or Endoscopic Nipple Sparing Mastectomy in the Management of Breast Cancer-Prospective Study
Acronym: RCENSM-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Intuitive Surgical (Industry); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCH-IRB-190414-P; 108-2314-B-371-006- (Other Grant/Funding Number: MOST)
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer Female
Keywords: nipple sparing mastectomy; robotic nipple sparing mastectomy (R-NSM); conventional nipple sparing mastectomy (C-NSM); endoscopic assisted nipple sparing mastectomy (E-NSM); immediate breast reconstruction (IBR); immediate prothesis breast reconstruction (IPBR)

STUDY DESIGN:
Intervention Model Description: prospective registry of R-NSM versus C-NSM or E-NSM in the management of breast cancer. 3 arms study for comparisons
Masking Description: prospective, non-randomized, non-masking, open label, 3 arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Robotic assisted nipple sparing mastectomy (R-NSM) (Experimental): R-NSM, which introduce da Vinci surgical platform through a small extra-mammary axillary or lateral chest wound to perform NSM.
  Interventions: Device: robotic assisted nipple sparing mastectomy
- Conventional nipple sparing mastectomy (C-NSM) (Active Comparator): Nipple-sparing mastectomy (NSM), which preserved the nipple areolar complex (NAC) and skin flap during mastectomy.
  Interventions: Procedure: Conventional nipple sparing mastectomy
- Endoscopic assisted nipple sparing mastectomy (E-NSM) (Active Comparator): E-NSM, which is performed through small axillary and/or peri-areolar incisions, with endoscopic instruments to performed nipple sparing mastectomy.
  Interventions: Procedure: Endoscopic assisted nipple sparing mastectomy

INTERVENTIONS:
Device: robotic assisted nipple sparing mastectomy — R-NSM, which introduce da Vinci surgical platform through a small extra-mammary axillary or lateral chest wound to perform NSM, had been applied in the surgical treatment of early breast cancer or risk reducing mastectomy. R-NSM, which incorporated 3-dimensional (3D) imaging system and flexibility of robotic arm and instruments, was reported to have the potential to overcome the technique difficulty of E-NSM.
  Arms: Robotic assisted nipple sparing mastectomy (R-NSM)
Procedure: Endoscopic assisted nipple sparing mastectomy — E-NSM, which is performed through small axillary and/or peri-areolar incisions, was reported to be associated with small inconspicuous incision and good cosmetic outcome. Conventional E-NSM was performed with two separate incisions over axilla and peri-areolar regions. E-NSM with areolar incision, just like NSM with areolar related incision (NAC ischemia/necrosis rate: range 7%-81.8%), was associated with increased NAC ischemia/necrosis (reported ranged: 9.1-19%). New technique modifications of E-NSM were emerging focusing on single axillary incision NSM, which spare the peri-areolar incision and thereby decrease the compromise of bloody supply from mastectomy skin flap, was reported to have low NAC necrosis rate (0%).
  Arms: Endoscopic assisted nipple sparing mastectomy (E-NSM)
Procedure: Conventional nipple sparing mastectomy — Nipple-sparing mastectomy (NSM), which preserved the nipple areolar complex (NAC) and skin flap during mastectomy, was increasingly performed in breast cancer patients due to better cosmetic outcome, higher patient satisfaction, and maintained oncologic safety.
  Arms: Conventional nipple sparing mastectomy (C-NSM)

SUMMARY:
This study will prospectively evaluate the surgical outcomes of robotic nipple sparing mastectomy (NSM) compared with endoscopic assisted NSM or conventional NSM in the management of breast cancer. One-third patients would received R-NSM, another one-third received C-NSM while the other one-third would receive E-NSM.

DETAILED DESCRIPTION:
Nipple-sparing mastectomy (NSM), which preserved the nipple areolar complex (NAC) and skin flap during mastectomy, was increasingly performed in breast cancer patients due to better cosmetic outcome, higher patient satisfaction, and maintained oncologic safety.

Minimal invasive surgery had become the main stream of operations, and new surgical innovations of NSM, like endoscopic nipple sparing mastectomy (E-NSM) or robotic nipple sparing mastectomy (R-NSM), were emerging and applied in the surgical treatment of breast cancer.

E-NSM, which is performed through small axillary and/or peri-areolar incisions, was reported to be associated with small inconspicuous incision and good cosmetic outcome. Conventional E-NSM was performed with two separate incisions over axilla and peri-areolar regions. E-NSM with areolar incision, just like NSM with areolar related incision (NAC ischemia/necrosis rate: range 7%-81.8%), was associated with increased NAC ischemia/necrosis (reported ranged: 9.1-19%). New technique modifications of E-NSM were emerging focusing on single axillary incision NSM, which spare the peri-areolar incision and thereby decrease the compromise of bloody supply from mastectomy skin flap, was reported to have low NAC necrosis rate (0%).

However, the 2-dimensional endoscopic in-line camera produces an inconsistent optical window around the curvature of the breast skin flap, and the internal mobility was limited and the dissection angles were inadequate with traditional endoscopic rigid tips instruments through single access. Due to the limitations of endoscopy instruments and technique difficulty, neither conventional E-NSM nor single access E-NSM was widespread used in breast cancer

R-NSM, which introduce da Vinci surgical platform through a small extra-mammary axillary or lateral chest wound to perform NSM, had been applied in the surgical treatment of early breast cancer or risk reducing mastectomy. R-NSM, which incorporated 3-dimensional (3D) imaging system and flexibility of robotic arm and instruments, was reported to have the potential to overcome the technique difficulty of E-NSM.

The preliminary results of R-NSM from current reported series and ours were safe, and associated with good cosmetic outcome and high patients' satisfaction. However, evidence comparing R-NSM to conventional NSM (C-NSM) or E-NSM was lacking.

In this study, the authors aim to investigate and analyze the clinical and aesthetic outcomes as well as the cost effectiveness of R-NSM through a prospective cohort of patients undergoing R-NSM, E-NSM or C-NSM.

ELIGIBILITY:
Inclusion Criteria:

* A. Indications and selection criteria for nipple sparing mastectomy (NSM) in general and conventional nipple sparing mastectomy (C-NSM)
* NSM will be offered to patients who are suitable for mastectomy but keen to conserve nipple areolar complex (NAC), with or without reconstruction. Patients must not have clinical or radiological involvement of the NAC. Patients with nipple involvement proven via intra-operative frozen section analysis will receive NAC excision and hence a skin-sparing mastectomy (SSM) performed instead.

B. Indications and selection criteria for robotic nipple sparing mastectomy (R-NSM) or endoscopic nipple sparing mastectomy (E-NSM)

* The general inclusion criteria or pre-requisite for nipple sparing mastectomy apply to R-NSM or E-NSM as well.
* In addition, R-NSM or E-NSM should only include early stage breast cancer (carcinoma in situ, stage I - IIIA), a tumor size less than 5 cm, no evidence of multiple lymph node metastasis, and no evidence of nipple, skin or chest wall invasion.

Exclusion Criteria:

* - Contraindications for R-NSM, C-NSM or E-NSM include those with apparent NAC involvement, inflammatory breast cancer, breast cancer with chest wall or skin invasion, locally advanced breast cancer, breast cancer with extensive axillary lymph node metastasis (stage III B or later), and patients with severe co-morbid conditions, such as heart disease, renal failure, liver dysfunction, and poor performance status as assessed by the primary physicians
* Relative contraindications include women with large (breast cup size larger than E or breast mastectomy weight >600gm) or ptotic breast as the aesthetic outcomes may be suboptimal.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Operation time | immediate post operation
  Overall operation time (minute), including breast cancer operations, lymph node surgery, and breast reconstructions
Morbidity and complications | within one month (30 days) post operation
  Delayed wound healing, degree of nipple ischemia/necrosis, seroma formation needing repeated aspiration, Blister formation, Skin flap ischemia necrosis, Hematoma formation, Implant loss will be collected and analyzed between different R-NSM, C-NSM and E-NSM groups.
Nipple areolar complex ischemia/necrosis grading | evaluated in post operative 2 weeks to 3 months post operation
  To evaluate the post-operative perfusion and survival of nipple areolar complex (NAC), a grading system was used in current study.
  The perfusion of NAC was evaluated in 2 weeks to 3 months post operation. The survival of NAC was confirmed at post-operative 3 months.
  The NAC ischemia/necrosis was divided into 5 different grades, which were:
  1. No ischemia/necrosis was observed in NAC (Grade I).
  2. Transient ischemia recovered without necrosis (Grade II).
  3. Partial ischemia/necrosis, recovered without loss of nipple volume (Grade III).
  4. Partial NAC necrosis with partial volume loss of nipple (Grade IV).
  5. Total NAC necrosis with all volume loss of nipple (Grade V). NAC ischemia/necrosis was segregated into no NAC necrosis (Grade I-III) and NAC necrosis (Grade IV-V).
  The ischemia/necrosis of NAC between different R-NSM, C-NSM and E-NSM groups were recorded and compared.
Surgical margin involvement | post operative 2 weeks after pathologic report available
  Surgical margin involvement was defined as tumor on the ink. The postoperative adjuvant hormone therapy, chemotherapy and radiotherapy were given to patients according to current breast cancer guidelines.
Aesthetic outcome evaluation-Patient reported cosmetic outcome results | 1-3 months after the operation when the wound was healed
  - Post-operative aesthetic results will be evaluated by comparing pre-operative and post-operative results. A self-reported questionnaire to evaluate the cosmetic outcome of breast cancer patients with mastectomy following breast reconstruction was conducted 1-3 months after the operation. This questionnaire comprises of 10 questions based on 4 itemized scales, which will be graded as "1, dis-satisfied", "2, fair", "3, satisfied", and "4, very satisfied".
Blood loss during operations | immediate post operation
  Blood loss (ml) from skin incision to completion of operations
Hospital stay | within 2 weeks of operation
  Hospital stay (days) during operation period, recorded from admission to day of discharge at the breast cancer operation.
Resection mastectomy weight | immediate post operation
  Mean mastectomy weight (gm) of patients received different mastectomy operations
Reconstruction implant volume | immediate post operation
  Reconstruction implant volume (ml)
Pain assessments | within post operation two weeks
  Pain assessments will also be collected as part of the post-operative parameters. Visual analogue scale (VAS) for pain assessments will be used in this study (range from 0 to 10 points, 0 indicate no pain, 10 indicate maximal pain ever experienced). VAS for pain per day would be recorded very day and compared.

SECONDARY OUTCOMES:
Cost- analysis of C-NSM versus R-NSM or E-NSM | post operation one month
  The medical cost associated with robotic versus conventional or endoscopic assisted NSM will be collected and compared. The medical cost incurred for each procedure include overall hospital cost. Information on surgery-related expenses will obtained from the finance department of the institution. In Taiwan, the operation fees of breast reconstruction and robotic breast surgery are not reimbursed by national insurance.
  * The medical cost covered by national insurance include operations fee for breast cancer and/or axillary lymph node surgery, anesthesia, admission fee, and all other medical related expenses.
  * The medical cost not reimbursed by national insurance, and needed to be paid for by patients include fees for breast reconstruction, robotic breast surgery, endoscopic breast surgery, instruments and prosthetic implants.
  * Cost is expressed in New Taiwan dollars (NTDs) and in United States dollars (USDs). An exchange rate of 31 NTD/USD was used to convert NTD to USD.
Disease free survival | 5 years post operation
  any local regional recurrence, or distant metastasis was recorded as an event. Disease free survival would be compared between R-NSM, C-NSM and E-NSM groups
Overall Survival | 5 years post operation
  overall survival would be compared between R-NSM, C-NSM and E-NSM groups

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Wen Lai, MD, PhD, Principal Investigator — Changhua Christian Hospital
Locations (11):
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung, Taiwan, Kaohsiung City
  - China Medical University Hospital, Taichung, Taiwan, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Shuang-Ho Hospital - Taipei Medical University, Taipei
  - Taipei Municipal Wan Fang Hospital, Tawian, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan, Taiwan, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petit JY, Veronesi U, Luini A, Orecchia R, Rey PC, Martella S, Didier F, De Lorenzi F, Rietjens M, Garusi C, Sonzogni A, Galimberti V, Leida E, Lazzari R, Giraldo A. When mastectomy becomes inevitable: the nipple-sparing approach. Breast. 2005 Dec;14(6):527-31. doi: 10.1016/j.breast.2005.08.028. Epub 2005 Oct 12. PMID 16226028
- [Background] Leff DR, Vashisht R, Yongue G, Keshtgar M, Yang GZ, Darzi A. Endoscopic breast surgery: where are we now and what might the future hold for video-assisted breast surgery? Breast Cancer Res Treat. 2011 Feb;125(3):607-25. doi: 10.1007/s10549-010-1258-4. Epub 2010 Dec 3. PMID 21128113
- [Background] Tukenmez M, Ozden BC, Agcaoglu O, Kecer M, Ozmen V, Muslumanoglu M, Igci A. Videoendoscopic single-port nipple-sparing mastectomy and immediate reconstruction. J Laparoendosc Adv Surg Tech A. 2014 Feb;24(2):77-82. doi: 10.1089/lap.2013.0172. Epub 2014 Jan 8. PMID 24401140
- [Background] Toesca A, Peradze N, Galimberti V, Manconi A, Intra M, Gentilini O, Sances D, Negri D, Veronesi G, Rietjens M, Zurrida S, Luini A, Veronesi U, Veronesi P. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction With Implant: First Report of Surgical Technique. Ann Surg. 2017 Aug;266(2):e28-e30. doi: 10.1097/SLA.0000000000001397. No abstract available. PMID 28692558
- [Background] Moran MS, Schnitt SJ, Giuliano AE, Harris JR, Khan SA, Horton J, Klimberg S, Chavez-MacGregor M, Freedman G, Houssami N, Johnson PL, Morrow M. Society of Surgical Oncology-American Society for Radiation Oncology consensus guideline on margins for breast-conserving surgery with whole-breast irradiation in stages I and II invasive breast cancer. Ann Surg Oncol. 2014 Mar;21(3):704-16. doi: 10.1245/s10434-014-3481-4. Epub 2014 Feb 10. PMID 24515565
- [Background] Park SW, Lee TJ, Kim EK, Eom JS. Managing necrosis of the nipple-areola complex in breast reconstruction after nipple-sparing mastectomy: immediate nipple-areola complex reconstruction with banked skin. Plast Reconstr Surg. 2014 Jan;133(1):73e-74e. doi: 10.1097/01.prs.0000436805.58165.d3. No abstract available. PMID 24374705
- [Result] Lai HW, Chen ST, Chen DR, Chen SL, Chang TW, Kuo SJ, Kuo YL, Hung CS. Current Trends in and Indications for Endoscopy-Assisted Breast Surgery for Breast Cancer: Results from a Six-Year Study Conducted by the Taiwan Endoscopic Breast Surgery Cooperative Group. PLoS One. 2016 Mar 7;11(3):e0150310. doi: 10.1371/journal.pone.0150310. eCollection 2016. PMID 26950469
- [Result] Lai HW, Lin SL, Chen ST, Kuok KM, Chen SL, Lin YL, Chen DR, Kuo SJ. Single-Axillary-Incision Endoscopic-Assisted Hybrid Technique for Nipple-Sparing Mastectomy: Technique, Preliminary Results, and Patient-Reported Cosmetic Outcome from Preliminary 50 Procedures. Ann Surg Oncol. 2018 May;25(5):1340-1349. doi: 10.1245/s10434-018-6383-z. Epub 2018 Feb 26. PMID 29484564
- [Result] Sakamoto N, Fukuma E, Higa K, Ozaki S, Sakamoto M, Abe S, Kurihara T, Tozaki M. Early results of an endoscopic nipple-sparing mastectomy for breast cancer. Ann Surg Oncol. 2009 Dec;16(12):3406-13. doi: 10.1245/s10434-009-0661-8. PMID 19662457
- [Result] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Result] Sarfati B, Struk S, Leymarie N, Honart JF, Alkhashnam H, Tran de Fremicourt K, Conversano A, Rimareix F, Simon M, Michiels S, Kolb F. Robotic Prophylactic Nipple-Sparing Mastectomy with Immediate Prosthetic Breast Reconstruction: A Prospective Study. Ann Surg Oncol. 2018 Sep;25(9):2579-2586. doi: 10.1245/s10434-018-6555-x. Epub 2018 Jun 29. PMID 29959612
- [Result] Lai HW, Chen ST, Lin SL, Chen CJ, Lin YL, Pai SH, Chen DR, Kuo SJ. Robotic Nipple-Sparing Mastectomy and Immediate Breast Reconstruction with Gel Implant: Technique, Preliminary Results and Patient-Reported Cosmetic Outcome. Ann Surg Oncol. 2019 Jan;26(1):42-52. doi: 10.1245/s10434-018-6704-2. Epub 2018 Aug 14. PMID 30109537
- [Result] Lai HW, Wang CC, Lai YC, Chen CJ, Lin SL, Chen ST, Lin YJ, Chen DR, Kuo SJ. The learning curve of robotic nipple sparing mastectomy for breast cancer: An analysis of consecutive 39 procedures with cumulative sum plot. Eur J Surg Oncol. 2019 Feb;45(2):125-133. doi: 10.1016/j.ejso.2018.09.021. Epub 2018 Oct 17. PMID 30360987
- [Result] Lai HW, Huang RH, Wu YT, Chen CJ, Chen ST, Lin YJ, Chen DR, Lee CW, Wu HK, Lin HY, Kuo SJ. Clinicopathologic factors related to surgical margin involvement, reoperation, and residual cancer in primary operable breast cancer - An analysis of 2050 patients. Eur J Surg Oncol. 2018 Nov;44(11):1725-1735. doi: 10.1016/j.ejso.2018.07.056. Epub 2018 Aug 1. PMID 30120037
- [Derived] Lai HW, Chen DR, Liu LC, Chen ST, Kuo YL, Lin SL, Wu YC, Huang TC, Hung CS, Lin YJ, Tseng HS, Mok CW, Cheng FT. Robotic Versus Conventional or Endoscopic-assisted Nipple-sparing Mastectomy and Immediate Prosthesis Breast Reconstruction in the Management of Breast Cancer: A Prospectively Designed Multicenter Trial Comparing Clinical Outcomes, Medical Cost, and Patient-reported Outcomes (RCENSM-P). Ann Surg. 2024 Jan 1;279(1):138-146. doi: 10.1097/SLA.0000000000005924. Epub 2023 May 25. PMID 37226826